CLINICAL TRIAL: NCT01293370
Title: Important Factors in Integration of Vocational Rehabilitation in Mental Health
Acronym: IVRMH
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: refKSH2910
Record Dates: First submitted 2011-01-21; First posted 2011-02-10 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Psychiatric Patients Experiences of Vocational Rehabilitation During Admittance in Hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- vocational rehabilitation: Admitted and discharged psychiatric patients receiving vocational rehabilitation

SUMMARY:
The purpose of this study is to explore, through a qualitative approach, how a group of people with serious mental illness experienced the integration of a vocational rehabilitation intervention during their admittance in hospital.

DETAILED DESCRIPTION:
People with serious mental illness admitted to hospital face significant barriers to gain both education and employment. Norway is a high-income welfare society with low unemployment rates, but the employment rates are very high in the population with psychosis and schizophrenia. Norway have a strategy for work and mental health, and through this strategy, the government has supported some pilot projects which focus on new ways of supporting people with serious mental illness in gaining employment. This study focuses on a representative sample participating in a pilot study. The sample consists of admitted patients who have received vocational rehabilitation under admittance. The study design is qualitative in nature with open- ended questions to allow the sample to express their opinions, attitudes and thoughts about the assistance they have had during their rehabilitation stay in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Formerly and present admitted patients in the Rehabilitation ward who participated in a project with vocational rehabilitation.

Exclusion Criteria:

* Mental retardation

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Admitted or discharged hospital patient, who also receives vocational rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Increase the understanding of the issues faced by people with serious mental illness who want to gain or maintain employment through vocational rehabilitation | From February 2011 - April 2011
  In order to explore the issues faced by people with serious mental illness in regard to maintain employment through vocational recovery, it was decided to use a qualitative approach. This approach was selected because it will give an understanding to a range of opinions and attitudes, and the reasons behind these attitudes through the use of open-ended questions. The primary outcome measure will be the range of opinions and attitudes that the representative sample provides.

SECONDARY OUTCOMES:
Identify the obstacles that people with serious mental illness face within the service delivery system on their pathway to gain employment | February 2011 - April 2011
  This study focus on a group of people with serious mental illness that have received a vocational rehabilitation intervention already while admitted to hospital. There is little research that focus on the integration of vocational rehabilitation given by vocational therapist during a hospital stay. With open-ended questions we will try to find out what this group of people think about the cooperation between different agencies on their pathway to recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Knut Sørgård, Dr.philos, Study Director — University of Northern Norway
Locations (1):
- Nordland Hospital trust, Bodø, Nordland County, Norway